CLINICAL TRIAL: NCT04633213
Title: A Phase 3, Multicenter, Randomized, Double-Blinded and Placebo-Controlled Study Evaluating the Efficacy and Safety of 0.25% HBM9036 (HL036) Ophthalmic Solution Compared to Placebo in Chinese Subjects With Moderate and Severe Dry Eye
Brief Title: A Study Evaluating HBM9036 Efficacy and Safety on Moderate to Severe Dry Eye
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9036.2
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2022-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBM9036 0.25% Ophthalmic Solution (Experimental): HBM9036, Ophthalmic Solution, twice a day, in the morning and evening
  Interventions: Drug: HBM9036 0.25% Ophthalmic Solution
- Placebo Ophthalmic Solution (Placebo Comparator): placebo, Ophthalmic Solution, twice a day, in the morning and evening
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HBM9036 0.25% Ophthalmic Solution — Ophthalmic Solution
  Arms: HBM9036 0.25% Ophthalmic Solution
Drug: Placebo — Ophthalmic Solution
  Arms: Placebo Ophthalmic Solution

SUMMARY:
The objective of this study is to compare the safety and efficacy of 0.25% HBM9036 (HL036) Ophthalmic Solution to placebo for the treatment of the Chinese subjects with moderate and severe dry eye.

DETAILED DESCRIPTION:
Inhibitors for tumor necrosis factor (TNF) have been widely used in clinical practice. Such class of medications have been approved for rheumatoid arthritis, ulcerative colitis, and uveitis. HBM9036 (HL036) is a molecularly engineered TNFR1 fragment, and molecule fragmentation and engineering techniques are applied for enhanced tissue distribution, increased stability and potency. In multiple early stage studies including preclinical studies, HBM9036 (HL036) has demonstrated the safety and efficacy in the therapy for moderate and severe dry eye. As a phase 3 confirmational study, this study is to evaluate the safety and efficacy of 0.25% HBM9036 (HL036) ophthalmic solution compared to placebo in Chinese subjects with moderate and severe dry eye.

ELIGIBILITY:
Inclusion Criteria:

1. At least 6 months history of any dry eye symptoms;
2. Must use or feel the need to use any types of eye drops to treat dry eye disease symptoms within 6 months prior to Screening Visit;
3. Best corrected visual acuity (BCVA) ≥ logMAR+0.7 as assessed according to the Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in both eyes at Screening Visit;
4. At least 1 eye dryness score ≥ 40mm measured by 100mm Visual Analogue Scale (VAS) at Screening Visit;
5. Schirmer's test score (anesthetized) ≥ 1mm and ≤ 10mm in the study eye at Screening Visit;
6. Average tear film breakup time (TFBUT) ≤5 seconds in the study eye at Screening Visit;
7. Total corneal fluorescein staining score ≥ 5.5 according to the Ora Calibra Corneal and Conjunctival Staining Scale at least in the study eye at Screening and Baseline Visits;
8. Conjunctival redness score ≥1 according to the Ora Calibra Conjunctival Redness Scale at least in the study eye at Screening Visit.

Exclusion Criteria:

1. At Screening Visit, Subjects observed by investigator with any clinically significant signs including active blepharitis and ocular allergies. Patients with meibomian gland dysfunction that need treatment;
2. Currently active ocular infection (bacterial, viral, or fungal) or any ocular surface inflammation;
3. Patients whose dry eye disease secondary to Sjogren's syndrome, Steven-Johnson Syndrome or chronic graft versus host disease, or patients suffered from serious autoimmune disorders such as systemic lupus erythematosus or rheumatoid arthritis, If their systemic disease are instable or drug application changed such as the type or dose of immunosuppressive biologics had been adjusted within 3 months or had drug withdrawal within 1 month or expected to have their drugs adjusted or discontinued during the study;
4. Planning to undergo any ocular or eyelid surgery;
5. Patients suffered from insertion of temporary lacrimal plug surgery within 6 months or insertion of permanent lacrimal plug surgery within 3 months. Or planning to undergo insertion of lacrimal plug surgery during the study;
6. Use of Cyclosporine A, Tacrolimus or Xiidra within 60 days prior to Screening Visit;
7. History of HBM9036 (HL036) use;
8. Currently use of prescription (including but not limited to antiglaucoma drops) or OTC drugs that locally applied to eyes, artificial tears, ophthalmic gel and eye rinse that cannot be interrupted during the study (excluding medications allowed in this study); pharmacological wash-out periods are required for some drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in total corneal staining scores (upper, central and lower cornea) of the study eye | 8 weeks
  Total corneal staining score (TCSS; superior, central, and inferior regions) of study eye evaluated by Ora Calibra® Corneal and Conjunctival Staining Scale for Grading of Fluorescein Staining at Visit 5/Day 57, change from baseline Score: From 0-12, a higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zuguo Liu, Doctor, Principal Investigator — Xiamen Eye Center Affiliated to Xiamen University
Locations (1):
- Xiamen Eye Center of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No